CLINICAL TRIAL: NCT03904576
Title: A Double-blind, Randomised, Two-way Cross-over, Single-dose, Placebo-controlled Trial to Investigate the Effects of BI 1358894 on Cholecystokinin Tetrapeptide (CCK-4) Induced Panic Symptoms in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test Whether BI 1358894 Reduces Druginduced Panic Symptoms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1402-0005; 2018-000057-41 (EudraCT Number)
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — TRPC inhibitor BI 1358894

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (T) (Experimental)
  Interventions: Drug: BI 1358894
- Reference Treatment (R) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1358894 — Film-coated tablet
  Arms: Treatment (T)
Drug: Placebo — Film-coated tablet
  Arms: Reference Treatment (R)

SUMMARY:
The main objective of this trial is to investigate the pharmacodynamic effects of a single dose of BI 1358894 on CCK-4- induced anxiogenic/ panic-like symptoms using the PSS in preselected CCK-4 sensitive healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Willingness to comply with contraception requirements. Subjects who are sexually active must use adequate contraception with their female partner throughout the study and until one month after the last administration of trial medication. Adequate methods are:

  * Sexual abstinence or
  * A vasectomy performed at least 1 year prior to screening (with medical assessment of the surgical success) or
  * Surgical sterilisation (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subject's female partner or
  * Postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with FSH above 40 U/L and estradiol below 30 ng/L is confirmatory) or
  * The use of condoms, if the female partner uses an adequate contraception method in addition, e.g., intrauterine device (IUD), hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first drug administration, or barrier method (e.g. diaphragm with spermicide)

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* C-Reactive Protein >ULN, erythrocyte sedimentation rate (ESR) ≥15 millimeters/h, liver or kidney parameter above ULN,
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication, CCK-4 or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 5 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Average intake of more than 21 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant Electrocardiogram (ECG) finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Any lifetime history of suicidal behaviour (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour)
* Any suicidal ideation of type 2 to 5 on the C-SSRS in the past 12 months (i.e. active suicidal thought, active suicidal thought with method, active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)
* Insufficient response to the CCK-4 challenge in Screening Visit 2

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- [Derived] Goettel M, Fuertig R, Mack SR, Just S, Sharma V, Wunder A, den Boer J. Effect of BI 1358894 on Cholecystokinin-Tetrapeptide (CCK-4)-Induced Anxiety, Panic Symptoms, and Stress Biomarkers: A Phase I Randomized Trial in Healthy Males. CNS Drugs. 2023 Dec;37(12):1099-1109. doi: 10.1007/s40263-023-01042-3. Epub 2023 Nov 29. PMID 38019356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A double-blind, randomized, two-way cross-over, single-dose, placebo-controlled trial to investigate the effects of BI 1358894 on cholecystokinin tetrapeptide (CCK-4) induced panic symptoms in healthy male subjects.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensure that all participants met all inclusion and non of the exclusion criteria. Participants were not to be entered to trial treatment in any of the specific entry criteria were not met.
Groups:
- 100 mg BI 1358894 (T) / Placebo (R): 4 film-coated tablets of 25 milligram (mg) of BI 1358894 were administered as a single oral dose with 240 milliliter (mL) of water after a standard high-fat meal as test treatment (T), followed by a washout period of at least 17 days, followed by 4 placebo film-coated tablets, administered as a single oral dose with 240 mL of water after a standard high-fat meal, as reference treatment (R). Treatments were administered 5 hours (h) prior to the provoking agent cholecystokinin tetrapeptide (CCK-4). CCK-4 was administered in 2 single doses of 50 microgram (μg) intravenous via bolus injection.
- Placebo (R) /100 mg BI 1358894 (T): 4 film-coated tablets of matching placebo were administered as a single oral dose with 240 milliliter (mL) of water after a standard high-fat meal as reference treatment (R), followed by a washout period of at least 17 days, followed by 4 film-coated tablets of 25 mg of BI 1358894, administered as a single oral dose with 240 mL of water after a standard high-fat meal, as test treatment (T). Treatments were administered 5 h prior to the provoking agent CCK-4. CCK-4 was administered in 2 single doses of 50 μg intravenous via bolus injection.
Period: Treatment Period 1
Arm/Group | 100 mg BI 1358894 (T) / Placebo (R) | Placebo (R) /100 mg BI 1358894 (T)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | 100 mg BI 1358894 (T) / Placebo (R) | Placebo (R) /100 mg BI 1358894 (T)
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1
Period: Treatment Period 2
Arm/Group | 100 mg BI 1358894 (T) / Placebo (R) | Placebo (R) /100 mg BI 1358894 (T)
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set: All participants that underwent screening procedures, entered the trial, and were documented to have received at least one dose of investigational study drug.
Groups:
- Placebo (R) / 100 mg BI 1358894 (T): 4 film-coated tablets of matching placebo were administered as a single oral dose with 240 milliliter (mL) of water after a standard high-fat meal as reference treatment (R), followed by a washout period of at least 17 days, followed by 4 film-coated tablets of 25 mg of BI 1358894, administered as a single oral dose with 240 mL of water after a standard high-fat meal, as test treatment (T). Treatments were administered 5 h prior to the provoking agent CCK-4. CCK-4 was administered in 2 single doses of 50 μg intravenous via bolus injection.
- Total: Total of all reporting groups
Arm/Group | 100 mg BI 1358894 (T) / Placebo (R) | Placebo (R) / 100 mg BI 1358894 (T) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.3 (10.0) | 27.0 (9.5) | 26.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 9 | 16
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Change From Baseline in Panic Symptom Scale (PSS) Sum Intensity Score
Description: The last value before administration of the CCK-4 challenge in each period was considered the corresponding period baseline measurement. The PSS sum intensity score mean value of the two period baseline values was considered as the subject baseline. The PSS is a patient reported outcome measurement from which the following factors where derived: physical symptoms of fear and the perception of alertness, anxiety, fear, and pain. The subjects were asked to rate each of 18 characteristic questions on a scale from 0 (absent) to 4 (very strong). The sum of the scale over all items constituted the PSS sum intensity score, ranging from 0 to 72. A higher score implies a stronger panic symptom.
Time Frame: Within 3 hours (h) prior trial medication administration and 4h, 4h 45 minutes (min), 5h 5min, 5h 10min, 5h 20min, 5h 30min and 192h thereafter.
Population: Pharmacodynamic set (PDS): All participants in the treated set (TS) who provided at least one primary pharmacodynamic parameter that was not excluded (due to protocol deviation or due to non-evaluability).
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- 100 mg BI 1358894 (T): 4 film-coated tablets of 25 milligram (mg) of BI 1358894 were orally administered with 240 milliliter (mL) of water after a standard high-fat meal as test treatment (T). The test treatment was administered 5 hours (h) prior to the provoking agent cholecystokinin tetrapeptide (CCK-4). 50 microgram (μg) CCK-4 were administered intravenous via bolus injection.
- Placebo (R): 4 film-coated tablets of matching placebo were orally administered with 240 milliliter (mL) of water after a standard high-fat meal as reference treatment (R).The reference treatment was administered 5 hours (h) prior to the provoking agent CCK-4. 50 μg CCK-4 were administered intravenous via bolus injection.
Arm/Group | 100 mg BI 1358894 (T) | Placebo (R)
Number analyzed (Participants) | 19 | 19
Score on a scale | 22.639 (2.880) | 29.944 (2.884)
Statistical Analysis 1: Comparison: 100 mg BI 1358894 (T) vs Placebo (R); Mixed effects model including effects for 'treatment', 'period' and 'subject' as well as covariates 'period baseline' and 'subject baseline'; Test type: Other; Difference of least squares means (T-R) = -7.305, 90% CI 2-sided [-10.949 to -3.661], Standard Error of Mean 2.082
Statistical Analysis 2: Comparison: 100 mg BI 1358894 (T) vs Placebo (R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Difference in % = -24.396 — Difference of least squares means in % (ratio to Placebo) (T-R)/R*100%

ADVERSE EVENTS:
Time Frame: From drug Administration until end of Trial, up to 40 days.
Description: Treated Set: All participants that underwent screening procedures, entered the trial, and were documented to have received at least one dose of investigational study drug.
Groups:
- 100 mg BI 1358894: 4 film-coated tablets of 25 milligram (mg) of BI 1358894 were orally administered with 240 milliliter (mL) of water after a standard high-fat meal as test treatment (T). The test treatment was administered 5 hours (h) prior to the provoking agent cholecystokinin tetrapeptide (CCK-4). 50 microgram (μg) CCK-4 were administered intravenous via bolus injection.
- Placebo: 4 film-coated tablets of matching placebo were orally administered with 240 milliliter (mL) of water after a standard high-fat meal as reference treatment (R).The reference treatment was administered 5 hours (h) prior to the provoking agent CCK-4. 50 μg CCK-4 were administered intravenous via bolus injection.
Arm/Group | 100 mg BI 1358894 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 14/19 | 10/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg BI 1358894 (N=19) | Placebo (N=19)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Catheter site induration (General disorders) | 0 | 1
Catheter site pain (General disorders) | 0 | 1
Catheter site paraesthesia (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 1
Feeling hot (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Medical device site irritation (General disorders) | 1 | 1
Vessel puncture site bruise (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 10 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Dissociative disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT03904576/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT03904576/SAP_001.pdf